CLINICAL TRIAL: NCT00263588
Title: A Phase II Study of Lapatinib for Brain Metastases in Subjects With ErbB2-Positive Breast Cancer Following Trastuzumab-based Systemic Therapy and Cranial Radiotherapy
Brief Title: Lapatinib for Brain Metastases In ErbB2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EGF105084; CLAP016A2202 (Other: Novartis); 2005-003944-68 (EudraCT Number)
Record Dates: First submitted 2005-12-02; First posted 2005-12-09 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Neoplasms, Breast
Keywords: breast cancer; brain metastases; ErbB2 positive; HER2 positive; neoplasms; cancer; lapatinib; LAP016A2202; LAP016A; CLAP016A2202; GW572016
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): 750 mg lapatinib administered orally twice daily
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — tyrosine kinase inhibitor

SUMMARY:
Determine how safe and effective lapatinib is when used to treat patients with ErbB2 overexpressing breast cancer that has spread to the brain and is still progressing there even after radiation treatment using WBRT (whole brain radiotherapy) or SRS (stereotactic radiosurgery) to the brain. Lapatinib is an oral drug that will be taken every day. Tests for safety and efficacy will be performed every 4 weeks or 8 weeks (depending on the test) during the course of the study.

ELIGIBILITY:
Inclusion criteria:

* Signed Informed Consent
* ErbB2(HER2)overexpressing breast cancer.
* Brain lesion(s) which are progressing.
* Prior treatment of brain metastases with Whole Brain Radiotherapy (WBR)and/or Stereotactic Radiosurgery (SRS).
* Prior treatment with trastuzumab (Herceptin), either alone or in combination with chemotherapy.
* Cardiac ejection fraction(LVEF)within the institutional range of normal as measured by Echocardiogram.
* Able to swallow an oral medication.
* Adequate kidney and liver function.
* Adequate bone marrow function.

Exclusion criteria:

* Pregnant or lactating females.
* Conditions that would effect the absorption of an oral drug.
* History of immediate or delayed hypersensitivity reaction to gadolinium contrast agents.
* Pre-existing severe cerebral vascular disease, such as stroke involving a major vessel.
* Serious medical or psychiatric disorder that would interfere with the patient's safety or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2005-12-02 (Actual); Primary Completion 2007-09-25 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- United States (25):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Sioux City, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Santa Fe, New Mexico
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Yakima, Washington
- Australia (7):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Ringwood East, Victoria
  - Novartis Investigative Site, Perth, Western Australia
  - Novartis Investigative Site, Adelaide
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Brussels, Belgium
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
- France (3):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
- Novartis Investigative Site, Neo Faliro, Greece
- India (2):
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Mumbai
- Italy (3):
  - Novartis Investigative Site, Reggio Emilia, Emilia-Romagna
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Perugia, Umbria
- Japan (3):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Tokyo
- Poland (2):
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Warsaw
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Uppsala, Sweden
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Locarno
- Taiwan (2):
  - Novartis Investigative Site, Tainan County
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Manchester, Lancashire
  - Novartis Investigative Site, Brighton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Sutherland S, Ashley S, Miles D, Chan S, Wardley A, Davidson N, Bhatti R, Shehata M, Nouras H, Camburn T, Johnston SR. Treatment of HER2-positive metastatic breast cancer with lapatinib and capecitabine in the lapatinib expanded access programme, including efficacy in brain metastases--the UK experience. Br J Cancer. 2010 Mar 16;102(6):995-1002. doi: 10.1038/sj.bjc.6605586. Epub 2010 Feb 23. PMID 20179708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Intent-to-Treat (ITT) Population: all subjects who received at least one dose of study medication
  Modified ITT (MITT) Population: all subjects who received at least four doses (750 mg lapatinib twice daily for two days) of study medication and who had measurable brain metastases (≥1 cm in diameter) at baseline assessment
Pre-assignment Details: Main phase: ITT 95 in Cohort A, 147 in Cohort B. MITT, 94 in Cohort A, and 143 subjects in Cohort B Optional open-label extension phase: 51 subjects. Long-term follow up (LTFU) Protocol amendment added on 15-Apr-2013
Groups:
- Cohort A: 750mg lapatinib administered orally twice daily. Cohort A subjects had Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and one or two prior trastuzumab-containing regimens, in total, for treatment of breast cancer in adjuvant and/or metastatic settings
- Cohort B: 750mg lapatinib administered orally twice daily. Cohort B subjects had ECOG performance status 2 and/or more than 2 prior trastuzumab-containing regimens for treatment of breast cancer in the adjuvant and/or metastatic settings.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 95 | 147
Completed | 14 | 15
Not Completed | 81 | 132
Not completed — Death | 54 | 90
Not completed — disease progression, coma, 1 unknown | 10 | 11
Not completed — Lost to Follow-up | 7 | 10
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Investigator decision | 7 | 15
Not completed — Sponsor terminated study | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population is defined as all subjects who received at least one dose of study medication.
Groups:
- Cohorts A: Overall - Main Study and Extension Phase - 750 mg lapatinib administered orally twice daily Cohort A subjects had Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and one or two prior trastuzumab-containing regimens, in total, for treatment of breast cancer in adjuvant and/or metastatic settings.
- Total: Total of all reporting groups
Arm/Group | Cohorts A | Cohort B | Total
Number analyzed (Participants) | 95 | 147 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] — Lapatinib Monotherapy - ITT Population
  years | 50.3 (10.33) | 49.3 (10.73) | 49.8 (10.53)
Age, Customized [Count of Participants; unit: Participants]
  <18 years: 242 | 0 | 0 | 0
  18-64 years: 242 | 85 | 135 | 220
  65-84 years: 242 | 10 | 11 | 21
  >85 years: 242 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 147 | 241
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African | 3 | 4 | 7
  American Indian/Alaskan Native | 0 | 1 | 1
  Asian - Central/South | 0 | 3 | 3
  Asian - Japanese | 6 | 0 | 6
  Asian - South-East Asian | 1 | 2 | 3
  Asia - East | 1 | 4 | 5
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African | 0 | 2 | 2
  White - White/ Caucasian/European | 83 | 129 | 212
  Mixed race | 0 | 1 | 1
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Central Nervous System (CNS) Best Overall Response
Description: Summary of CNS Objective Response (Lapatinib Monotherapy - MITT Population)
  Response to lapatinib in patients with progressive brain metastases from ErbB2-overexpressing breast cancer.
  The primary indicator of drug efficacy was CNS objective response rate. A CNS objective response was defined as either a Complete response (CR) or Partial response (PR), as assessed by volumetric analysis of brain Magnetic resonance imaging (MRI), provided there was no progression of systemic disease outside of the CNS, increasing steroid requirements, or worsening of Neurological signs and symptoms (NSS)
  A CNS objective response rate was defined as a 50% volumetric reduction in sum of CNS target lesions, with no new or progressive CNS or non-CNS lesions, no increases in tumor-related steroid requirements and no worsening of neurological signs or symptoms
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: Modified ITT (MITT) Population is defined as all subjects who received at least four doses (750 mg lapatinib 2x daily for 2 days) of study medication and who had measurable brain metastases (greater than or equal to 1cm in diameter) at baseline assessment. MITT was the primary population for analysis of efficacy data in lapatinib monotherapy arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 6 | 9
  Stable disease (SD) | 40 | 46
  Progressive disease (PD) | 40 | 70
  Unknown | 8 | 18

2. Primary Outcome: The Percentage of Participants With Central Nervous System (CNS) Objective Response Rate - Response Rate (CR + PR)
Description: Summary of CNS Objective Response (the Complete Response + Partial Response)
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
percentage of participants | 6 [2.4 to 13.4] | 6 [2.9 to 11.6]

3. Secondary Outcome: Percentage of Participants With Improvement in Neurological Signs and Symptoms (NSS) Measured Using the Neurological Examination Worksheet
Description: Physician-reported NSS worksheet is derived from 13 AEs and measured by NCI CTCAE v3.0 grouped into 7 categories: level of consciousness, neurological symptoms, cranial nerves, language, strength, sensation, & ataxia. Improvement of NSS required: Decrease by 1 or more grades from baseline of any tumor-related NSS, with confirmation at least 4 wks later, No development or worsening in any tumor-related NSS during interval, No radiographic evidence of CNS progression (assessed by volumetric MRI) or systemic (non-CNS) progression (assessed by RECIST) during interval, Stable or decreasing steroids during interval as defined by GSK equivalent doses of an alternative corticosteroid or a dose increase for non-tumor related reasons didn't constitute a steroid increase. Improvement in any non-tumor associated NSS didn't constitute improvement in NSS. Neurological exam, using Neurological Examination Worksheet was assessed at baseline & each 4 wks. Categories below are not mutually exclusive.
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: MITT population
  Analysis was performed on combined cohorts in order to have a sufficient sample size to analyze association of CNS Volumetric Change from Baseline and NSS Improvement
Measure: Count of Participants; unit: Participants
Groups:
- Cohorts A and B: Overall - Main Study and Extension Phase - 750 mg lapatinib administered orally twice daily
Arm/Group | Cohorts A and B
Number analyzed (Participants) | 237
Participants
  Subjects with NSS improvement: number analyzed (Participants) | 198
  Subjects with NSS improvement | 24
  >=20% volumetric reduction of lesion: number analyzed (Participants) | 34
  >=20% volumetric reduction of lesion | 8
  any volumetric reduction of lesion: number analyzed (Participants) | 59
  any volumetric reduction of lesion | 14
  volumetric increase or withdrew: number analyzed (Participants) | 125
  volumetric increase or withdrew | 9

4. Secondary Outcome: Percentage of Subjects With a CNS Objective Response or Improvement in Baseline Neurological Signs and Symptoms (NSS)
Description: Summary of Proportion of Subjects with a CNS Objective Response or Improvement in Baseline NSS
Time Frame: baseline and weeks 8, 16, 24, 32, 40, 48
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
percentage of participants
  week 8: number analyzed (Participants) | 79 | 110
  week 8 | 23 [14.1 to 33.6] | 14 [7.8 to 21.5]
  week 16: number analyzed (Participants) | 43 | 50
  week 16 | 2 [0.1 to 12.3] | 8 [2.2 to 19.2]
  week 24: number analyzed (Participants) | 12 | 19
  week 24 | 8 [0.2 to 38.5] | 11 [1.3 to 33.1]
  week 32: number analyzed (Participants) | 6 | 3
  week 32 | 17 [0.4 to 64.1] | 0.0 [0.0 to 0.0]
  week 40: number analyzed (Participants) | 3 | 2
  week 40 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  week 48: number analyzed (Participants) | 2 | 2
  week 48 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

5. Secondary Outcome: Duration of Central Nervous System (CNS) Objective Response
Description: The duration of CNS objective response, defined as the time from first CNS
  Objective response until tumor progression at any site or death due to any cause.
  A CNS objective response was defined as either a Complete Response (CR) or Partial Response (PR), as assessed by volumetric analysis of magnetic resonance imaging (MRI), provided there was no progression of systemic disease outside of the CNS, increasing steroid requirements, or worsening of tumor-related neurological signs or symptoms.
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: Lapatinib monotherapy MITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
months | 2.43 [0.99 to NA] — Upper limit Not evaluable (Due to the low number of CNS responders, a meaningful interpretation of duration of response is not possible). | 1.58 [0.99 to 3.55]

6. Secondary Outcome: Percentage of Patients With CNS Disease Control (Complete Response, Partial Response or Stable Disease) at 6 Months of Lapatinib Therapy
Description: The CNS disease control rate, defined as the percentage of subjects with CR, PR or stable disease at Week 24
Time Frame: from Start of lapatinib to 6 months
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
percentage of participants | 9 [3.7 to 16.1] | 2 [0.4 to 6.0]

7. Secondary Outcome: Time to Progression (TTP) at Any Site
Description: Summary of Kaplan-Meier Estimates for Progression Free Survival at Any Site
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: Lapatinib Monotherapy MITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
months | 2.60 [1.87 to 3.25] | 1.87 [1.84 to 2.63]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from initiation of investigational product to death due to any cause.
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: Lapatinib Monotherapy MITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
months | 10.78 [7.95 to 12.68] | 5.82 [4.78 to 7.89]

9. Secondary Outcome: Summary of Site of First Progression
Description: baseline to time of disease progression or death
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 94 | 143
Participants
  CNS progression | 69 | 72
  Non-CNS prgression | 1 | 10
  CNS and Non-CNS progression | 12 | 36

10. Secondary Outcome: Primary Cause of Death
Description: Summary of Overall All-cause mortality (Main Study and Extension)
Time Frame: time from baseline to data cutoff (25 Sept 2007); approximately 2 years
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 95 | 147
Participants
  Disease under study | 74 | 124
  Other | 4 | 4

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 12 months.
Description: All cause mortality (on-treatment deaths) was collected for as long as participants could be contacted from FPFV until LPLV up to a maximum of 12 years and 3 months
  SAEs are presented from main and extension phase
Groups:
- EGF105084/Cohort A: Cohort A subjects had Eastern Cooperative Oncology Group (ECOG) performance status 0-1, and one or two prior trastuzumab-containing regimens, in total, for treatment of breast cancer in adjuvant and/or metastatic settings
- EGF105084/Cohort B: Cohort B subjects had ECOG performance status 2 and/or more than 2 prior trastuzumab-containing regimens for treatment of breast cancer in the adjuvant and/or metastatic settings
Arm/Group | EGF105084/Cohort A | EGF105084/Cohort B
All-Cause Mortality (participants affected / at risk) | 78/95 | 128/147
Serious Adverse Events (participants affected / at risk) | 36/95 | 52/147
Other Adverse Events (participants affected / at risk) | 90/95 | 131/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGF105084/Cohort A (N=95) | EGF105084/Cohort B (N=147)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 5
Asthenia (General disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 3
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 5
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
On treatment deaths (General disorders) | 20 | 48 — All participants who died while on treatment of all disorders
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EGF105084/Cohort A (N=95) | EGF105084/Cohort B (N=147)
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 9 | 16
Diarrhoea (Gastrointestinal disorders) | 71 | 92
Dry mouth (Gastrointestinal disorders) | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 9
Nausea (Gastrointestinal disorders) | 29 | 47
Vomiting (Gastrointestinal disorders) | 24 | 39
Asthenia (General disorders) | 9 | 15
Fatigue (General disorders) | 30 | 29
Oedema peripheral (General disorders) | 6 | 16
Pyrexia (General disorders) | 5 | 6
Nasopharyngitis (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 7 | 8
Alanine aminotransferase increased (Investigations) | 4 | 13
Blood bilirubin increased (Investigations) | 7 | 1
Weight decreased (Investigations) | 5 | 11
Decreased appetite (Metabolism and nutrition disorders) | 16 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 7
Dizziness (Nervous system disorders) | 8 | 5
Dysgeusia (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 24 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Acne (Skin and subcutaneous tissue disorders) | 6 | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 13
Rash (Skin and subcutaneous tissue disorders) | 40 | 37

LIMITATIONS AND CAVEATS:
Outcome Quantitative Toxicities Associated with Oral Lapatinib are in Adverse Events section. No analysis was performed for 2 outcomes: Relationship of PET Uptake, as Predictors of Response; and Relationship Between Genetic Variants in Select Genes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e.; data from all sites) in the clinical trial.